CLINICAL TRIAL: NCT03180034
Title: A Scientific Evaluation of One or Two Doses of Vaccine Against Human Papillomavirus: the ESCUDDO Study ("Estudio de Comparacion de Una y Dos Dosis de Vacunas Contra el Virus de Papiloma Humano (VPH)")
Brief Title: Comparing One or Two Doses of the Human Papillomavirus Vaccine for the Prevention of Human Papillomavirus Infection, ESCUDDO Study
Acronym: ESCUDDO
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Collaborators: Bill and Melinda Gates Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: NCI-2020-08550; NCI-2020-08550 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CEC-HCB-E006-2024; 17-C-N108 (Other: National Cancer Institute)
Record Dates: First submitted 2017-06-07; First posted 2017-06-08 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-09

CONDITIONS: Human Papillomavirus Infection; Human Papillomavirus-Related Cervical Carcinoma
MeSH Terms: conditions — Papillomavirus Infections | interventions — Diphtheria Toxoid; adacel; Diphtheria-Tetanus-acellular Pertussis Vaccines; Tetanus Toxoid; human papillomavirus vaccine, L1 type 16, 18; Human Papillomavirus Recombinant Vaccine nonavalent

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Specimen lab
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Arm I (Gardasil, Tdap) (Experimental): Participants receive Gardasil IM at month 0 and Tdap IM at month 6.
  Interventions: Biological: Diphtheria Toxoid/Tetanus Toxoid/Acellular Pertussis Vaccine Adsorbed; Other: Questionnaire Administration; Biological: Recombinant Human Papillomavirus Nonavalent Vaccine
- Arm II (Cervarix, Tdap) (Experimental): Participants receive Cervarix IM at month 0 and Tdap IM at month 6.
  Interventions: Biological: Diphtheria Toxoid/Tetanus Toxoid/Acellular Pertussis Vaccine Adsorbed; Other: Questionnaire Administration; Biological: Recombinant Human Papillomavirus Bivalent Vaccine
- Arm III (Gardasil) (Active Comparator): Participants receive Gardasil IM at month 0 and 6.
  Interventions: Other: Questionnaire Administration; Biological: Recombinant Human Papillomavirus Nonavalent Vaccine
- Arm IV (Cervarix) (Active Comparator): Participants receive Cervarix IM at month 0 and 6.
  Interventions: Other: Questionnaire Administration; Biological: Recombinant Human Papillomavirus Bivalent Vaccine
- Arm V (epidemiologic survey) (No Intervention): A concurrent epidemiologic survey for HPV status among two groups of unvaccinated women. Survey participants are followed for two study visits six months apart to determine their HPV DNA status, with no further follow-up. These women will be offered HPV vaccination (Cervarix) at the two study visits.

INTERVENTIONS:
Biological: Diphtheria Toxoid/Tetanus Toxoid/Acellular Pertussis Vaccine Adsorbed — Given IM
  Other Names: Adacel; Daptacel; Diphtheria and Tetanus Toxoids and Acellular Pertussis Vaccine Adsorbed; Diphtheria Toxoid Tetanus Toxoid Acellular Pertussis Vaccine Adsorbed; Diphtheria Toxoid/Tetanus Toxoid/Acellular Pertussis Vaccine; DTaP; Infanrix; Tripedia
  Arms: Arm I (Gardasil, Tdap); Arm II (Cervarix, Tdap)
Other: Questionnaire Administration — Ancillary studies
  Arms: Arm I (Gardasil, Tdap); Arm II (Cervarix, Tdap); Arm III (Gardasil); Arm IV (Cervarix)
Biological: Recombinant Human Papillomavirus Bivalent Vaccine — Given IM
  Other Names: Cervarix; GSK-580299; HPV 16/18 L1 VLP/AS04 VAC; HPV-16/18 VLP/AS04 Vaccine; Human Papillomavirus 16/18 L1 Virus-Like Particle/AS04 Vaccine; Human Papillomavirus Bivalent Types 16 and 18 Vaccine, Recombinant; Human Papillomavirus Vaccine L1 16,18; Human Papillomavirus Vaccine, L1 Type 16, 18; Recombinant HPV Bivalent Vaccine
  Arms: Arm II (Cervarix, Tdap); Arm IV (Cervarix)
Biological: Recombinant Human Papillomavirus Nonavalent Vaccine — Given IM
  Other Names: Gardasil 9; Nonavalent HPV VLP Vaccine; Recombinant HPV Nonavalent Vaccine; Recombinant Human Papillomavirus 9-valent Vaccine
  Arms: Arm I (Gardasil, Tdap); Arm III (Gardasil)

SUMMARY:
This phase IV trial investigates whether one dose of a human papillomavirus vaccine works as well as two doses in preventing human papillomavirus (HPV) infection. Certain types of HPV cause almost all cases of cervical cancer. Vaccines that protect against infection with these types of human papillomavirus may reduce the risk of cervical cancer. Both Gardasil-9 and Cervarix protect against HPV 16 and 18, which cause 70% of all cervical cancers. However, HPV vaccination rates are too low, especially in countries with very high rates of cervical cancer. HPV vaccines are expensive-many countries cannot afford them-more than one dose is needed, and giving multiple doses is difficult. Researchers want to find out if one dose prevents HPV infection. If it does, more people might get the vaccine.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. For each vaccine separately, to evaluate non-inferiority of one compared to two vaccination doses in the prevention of new HPV16/18 cervical HPV infections that persist 6+ months in girls ages 12-16 years at vaccination.

II. For each vaccine separately, to evaluate one dose of HPV vaccination compared to no vaccination in the protection against HPV16/18 cervical HPV infections that persist 6+ months in girls ages 12-16 years at vaccination; protection resultant from two HPV vaccine doses compared to no vaccination will also be investigated. Note that the second epidemiological survey group (the end-of-study survey or EOSS) will serve as the primary unvaccinated group for these analyses.

SECONDARY OBJECTIVES:

I. For each vaccine separately, to compare immunogenicity via measurement of serum antibodies between girls who received one and two doses of the HPV vaccines. When looking at these antibodies, the primary focus will be on HPV16/18; antibodies against additional HPV types included in the nonavalent HPV vaccine will also be investigated.

II. For each vaccine separately, estimate (a) infection rate difference of one versus two doses, and (b) one-dose VE compared to no vaccination and (c) two-dose VE compared to no vaccination, in the following groupings of cervical HPV infections that persists 6+ months:

IIa. 12 carcinogenic HPV types (16/18/31/33/35/39/45/51/52/56/58/59, aggregated); IIb. 10 carcinogenic HPV types excluding 16/18 (31/33/35/39/45/51/52/56/58/59, aggregated); IIc. 7 carcinogenic HPV types included in the nonavalent HPV vaccine formulation (16/18/31/33/45/52/58, aggregated); IId. HPV types cCross-protected by the ASO-4 adjuvanted bivalent vaccine (31/33/45, aggregated); IIe. Each of the carcinogenic types (16/18/31/33/35/39/45/51/52/56/58/59, individually); IIf. 2 non-carcinogenic, genital warts-associated HPV types (6/11, aggregated). III. For the nonavalent vaccine, investigate non-inferiority of one compared to two vaccination doses in the prevention of cervical HPV infections that persist 6+ months compared to a pre-specified bound. for the 7 carcinogenic HPV types protected by the nonavalent vaccine (16/18/31/33/45/52/58, aggregated).

ANCILLARY OBJECTIVES:

I. Conduct a cost and cost-effectiveness evaluation of HPV vaccination with one versus two doses of the nonavalent and bivalent vaccines in the setting of Costa Rica (See complementary study protocol entitled: Complementary micro-costing and cost- effectiveness study for the clinical trial: "A scientific evaluation of one and two doses of the bivalent and nonavalent prophylactic HPV vaccines").

II. To perform an evaluation of each vaccine at 4 years. IIa. For each vaccine separately, evaluate non-inferiority of one compared to two vaccination doses in the prevention of new HPV16/18 cervical HPV infections that persist 6+ months in girls ages 12-16 years at vaccination using the first four years of data; IIb. For each vaccine separately, evaluate one dose of HPV vaccination compared to no vaccination in the protection against HPV16/18 cervical HPV infections that persist 6+ months in girls ages 12-16 years at vaccination using data available at four years and the first epidemiologic survey; protection resultant from two doses of the HPV vaccines compared to no vaccination will also be investigated.

III. For each vaccine separately, calculate the infection rate difference of one versus two doses, and vaccine efficacy, for the following study endpoints (including but not limited to those listed below):

IIIa. Any new HPV16, HPV18, or HPV16/18 infection (i.e., one-time detection); IIIb. Any new carcinogenic-type HPV infection (i.e., one-time HPV detection of aggregate HPV vaccine and/or non-vaccine HPV types); IIIc. Any new vaccine-type HPV infection (i.e., aggregate HPV 16/18/31/33/45/52/58); IIId. Any new HPV6/11 infection (i.e., one-time detection). IV. Compare HPV attack rate and immunogenicity of Merck nonavalent versus (vs.) GlaxoSmithKline (GSK) bivalent vaccines with respect to number of vaccine doses received in the prevention of six-month persistent HPV16/18 and any carcinogenic infections, and in the prevention of one-time detection of these types.

V. Conditional on demonstrating inferiority of one versus two doses of the vaccine (Primary Objective #1), to evaluate A) inferiority of one versus two doses and B) reduction in the HPV attack rate of one and two doses compared to none by time (years 1 through 4).

VI. Obtain participants authorization to passively track cervical pre-cancer, carcinoma in situ and cervical cancer outcomes through the national tumor registry, national cytology laboratory, social security registries, national cytology laboratory, and other resources after the trial ends (i.e., to continue indefinitely or until consent is rescinded).

VII. Establish a biobank including blood components (for example but not limited to serum, red blood cells, plasma, peripheral blood mononuclear cells), urine, oral and cervical swab samples collected from girls in the randomized trial and the epidemiologic HPV survey for futures analysis related to HPV infection, associated diseases, and effects of the vaccine.

OUTLINE: There are two components to the study: (1) a controlled, randomized, double-blinded non-inferiority clinical trial to compare one-dose to two-dose vaccination among twenty thousand girls 12 to 16 years old; and (2) an epidemiologic survey for HPV status among unvaccinated women 16-21 years old, enrolled concurrent with the final two visits of the trial to serve as the unvaccinated group. Trial participants are randomized to 1 of 4 arms. Survey participants are assigned to Arm V.

ARM I: Participants receive recombinant human papillomavirus nonavalent vaccine (Gardasil) intramuscularly (IM) at month 0 and diphtheria toxoid/tetanus toxoid/acellular pertussis vaccine adsorbed (Tdap) IM at month 6.

ARM II: Participants receive recombinant human papillomavirus bivalent vaccine (Cervarix) IM at month 0 and Tdap IM at month 6.

ARM III: Participants receive Gardasil IM at month 0 and 6.

ARM IV: Participants receive Cervarix IM at month 0 and 6.

After completion of study intervention, trial participants are followed up every 6 months for up to 4 years.

ARM V: A concurrent epidemiologic survey for HPV status among two groups of unvaccinated women. Survey participants are followed for two study visits six months apart to determine their HPV deoxyribonucleic acid (DNA) status, with no further follow-up. These women will be offered HPV vaccination (Cervarix) at the two study visits.

ELIGIBILITY:
Inclusion Criteria:

* RANDOMIZED TRIAL ELIGIBILITY CRITERIA: Female
* RANDOMIZED TRIAL ELIGIBILITY CRITERIA: Aged between 12 and 16 years inclusive
* RANDOMIZED TRIAL ELIGIBILITY CRITERIA: Living in the study area without plans to move outside the country in the next six months
* RANDOMIZED TRIAL ELIGIBILITY CRITERIA: Able to communicate with study personnel
* RANDOMIZED TRIAL ELIGIBILITY CRITERIA: Willing to participate in the study and sign the informed assent
* RANDOMIZED TRIAL ELIGIBILITY CRITERIA: Supported in study participation by at least one of their parents (or guardians), who is willing to sign the informed consent document
* RANDOMIZED TRIAL ELIGIBILITY CRITERIA: In good health as determined by a medical history (physical exam will be conducted if necessary per the doctor's criterion)
* INITIAL SURVEY ELIGIBILITY CRITERIA: Same as trial participants except for the age range, which is between 17 and 20 years old inclusive
* END-OF-STUDY SURVEY ELIGIBILITY CRITERIA: Same as trial and initial survey participants except for the age range, which will be closely matched to the current ages of trial participants when they are attending their E54 visits, and thus is expected to be approximately between 16 and 21 years old inclusive

Exclusion Criteria:

* RANDOMIZED TRIAL ELIGIBILITY CRITERIA: They have a diagnosis of an autoimmune, degenerative, or neurological disease without treatment or adequate control; a progressive or severe neurological disease; a genetic immunodeficiency; or any other serious chronic disease without treatment and / or adequate control that, according to the principal investigator or designee, for which vaccination is contraindicated (NOTE: Potential participants with these conditions can be included after consultation with the external medical advisor of the study or with an appropriate specialist
* RANDOMIZED TRIAL ELIGIBILITY CRITERIA: They are allergic to one of the vaccine components, yeast, or latex
* RANDOMIZED TRIAL ELIGIBILITY CRITERIA: The clinician determining the eligibility in agreement with principal investigator considers that there is a reason that precludes participation
* RANDOMIZED TRIAL ELIGIBILITY CRITERIA: They have been vaccinated against HPV
* RANDOMIZED TRIAL ELIGIBILITY CRITERIA: The girl or her parent/legal guardian does not have an identification document
* INITIAL SURVEY ELIGIBILITY CRITERIA: Same as trial participants
* END-OF-STUDY SURVEY ELIGIBILITY CRITERIA: They have a positive or equivocal urine pregnancy test result
* END-OF-STUDY SURVEY ELIGIBILITY CRITERIA: They are pregnant
* END-OF-STUDY SURVEY ELIGIBILITY CRITERIA: investigator considers that there is a reason that precludes participation
* END-OF-STUDY SURVEY ELIGIBILITY CRITERIA: They have been vaccinated against HPV
* END-OF-STUDY SURVEY ELIGIBILITY CRITERIA: They or their parent/legal guardian, as applicable, does not have an identification document

Ages: 12 Years to 21 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 27945 (Actual)
Dates: Start 2017-11-29 (Actual); Primary Completion 2025-08-21 (Actual); Study Completion 2028-08-01 (Estimated)

PRIMARY OUTCOMES:
Occurrence of at least one incident persistent human papillomavirus (HPV)-16 and/or HPV-18 cervical infections, counted cumulatively over the follow-up visits | Months 12 to 60
  To be considered incident and persistent, an HPV-16 and/or HPV-18 infection must fulfill the following criteria: Two same-type HPV positive (by polymerase chain reaction [PCR]) test results 3+ months apart at consecutive study visits reported after the 6-month visit (i.e. 12-month visit or later); type-specific HPV negative results from baseline and 6 month visits.
Incident persistent HPV-16 and/or HPV-18 cervical infections | Months 54 and 60
  Same type infection at 54 and 60-month visits, and absence of infection at the both 0- and 6-month visits.
Persistent HPV-16 and/or HPV-18 cervical infections (End-of-Study Survey Cohort) | Baseline, and 6 months

SECONDARY OUTCOMES:
HPV-16 and HPV-18 antibody concentration based on the Luminex bead-based multiplex immunoassay (LIA) assay | Up to 36 months
  Will be obtained from blood specimens (serum). To confirm that HPV-16 and HPV-18 LIA results reflect neutralization potential, the HPV-16 and HPV- 18 neutralization assays will also be evaluated on a subset of individuals (30 per arm * 4 arms * 9 visits * 2 assays = 2160 assays) and correlated with the LIA results.
Incident-persistent HPV infections, defined similarly as the primary outcomes, but in different groupings of HPV types | Months 12 to 60
  * 12 carcinogenic HPV types (16/18/31/33/35/39/45/51/52/56/58/59, aggregated)
  * 10 carcinogenic HPV types excluding 16/18 (31/33/35/39/45/51/52/56/58/59, aggregated)
  * 7 carcinogenic HPV types included in the nonavalent HPV vaccine (16/18/31/33/45/52/58, aggregated)
  * HPV types cross-protected by the ASO-4 adjuvanted bivalent vaccine (31/33/45, aggregated)
  * Each of the carcinogenic types (16/18/31/33/35/39/45/51/52/56/58/59, individually)
  * 2 non-carcinogenic genital warts-associated HPV types (6/11, aggregated)

CONTACTS AND LOCATIONS:
Overall Officials: Aimee R Kreimer, Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- Agencia Costarricense de Investigaciones Biomédicas (ACIB), Liberia, Guanacaste Province, Costa Rica

REFERENCES:
- [Derived] Kreimer AR, Porras C, Liu D, Hildesheim A, Carvajal LJ, Ocampo R, Romero B, Gail MH, Cortes B, Sierra MS, Coronado K, Sampson J, Coto C, Dagnall CL, Mora D, Kemp TJ, Zuniga M, Pinto LA, Barrientos G, Schussler J, Estrada Y, Montero C, Avila C, Ruggieri D, Cyr JT, Chanock S, Lowy DR, Schiller JT, Herrero R. Noninferiority of One HPV Vaccine Dose to Two Doses. N Engl J Med. 2025 Dec 18;393(24):2421-2433. doi: 10.1056/NEJMoa2506765. Epub 2025 Dec 3. PMID 41337735
- [Derived] Bergman H, Henschke N, Arevalo-Rodriguez I, Buckley BS, Crosbie EJ, Davies JC, Dwan K, Golder SP, Loke YK, Probyn K, Petkovic J, Villanueva G, Morrison J. Human papillomavirus (HPV) vaccination for the prevention of cervical cancer and other HPV-related diseases: a network meta-analysis. Cochrane Database Syst Rev. 2025 Nov 24;11(11):CD015364. doi: 10.1002/14651858.CD015364.pub2. PMID 41276263
- [Derived] Porras C, Sampson JN, Herrero R, Gail MH, Cortes B, Hildesheim A, Cyr J, Romero B, Schiller JT, Montero C, Pinto LA, Schussler J, Coronado K, Sierra MS, Kim JJ, Torres CM, Carvajal L, Wagner S, Campos NG, Ocampo R, Kemp TJ, Zuniga M, Lowy DR, Avila C, Chanock S, Castrillo A, Estrada Y, Barrientos G, Monge C, Oconitrillo MY, Kreimer AR. Rationale and design of a double-blind randomized non-inferiority clinical trial to evaluate one or two doses of vaccine against human papillomavirus including an epidemiologic survey to estimate vaccine efficacy: The Costa Rica ESCUDDO trial. Vaccine. 2022 Jan 3;40(1):76-88. doi: 10.1016/j.vaccine.2021.11.041. Epub 2021 Nov 29. PMID 34857420
- [Derived] Teppler H, Bautista O; Thomas Group; Flores S, McCauley J, Luxembourg A. Design of a Phase III immunogenicity and safety study evaluating two-dose regimens of 9-valent human papillomavirus (9vHPV) vaccine with extended dosing intervals. Contemp Clin Trials. 2021 Jun;105:106403. doi: 10.1016/j.cct.2021.106403. Epub 2021 Apr 12. PMID 33857679
- [Derived] Kreimer AR, Cernuschi T, Rees H, Saslow D, Porras C, Schiller J. Prioritisation of the human papillomavirus vaccine in a time of constrained supply. Lancet Child Adolesc Health. 2020 May;4(5):349-351. doi: 10.1016/S2352-4642(20)30038-9. Epub 2020 Feb 17. No abstract available. PMID 32078808